CLINICAL TRIAL: NCT05342506
Title: A Open, Single Arm, Phase IIa Clinical Study on the Safety, Pharmacokinetics, and Efficacy of ScTIL (Genetically Modified Tumor Infiltrating Lymphocytes) in the Treatment of Gynecological Malignancies
Brief Title: Clinical Study on the Safety, Pharmacokinetics, and Efficacy of ScTIL (Genetically Modified Tumor Infiltrating Lymphocytes) in the Treatment of Gynecological Malignancies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Chineo Medicine (Beijing) Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHKT-SCT006-2022
Record Dates: First submitted 2022-03-09; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-03

CONDITIONS: Cervical Cancer; Ovarian Cancer; Malignant Trophoblastic Tumor
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Study subjects: Patient with cervical carcinoma
  Interventions: Drug: Toripalimab + ScTIL
- Cohort 2 (Experimental): Study subjects: Patient with ovarian cancer
  Interventions: Drug: Toripalimab + ScTIL
- Cohort 3 (Experimental): Study subjects: Patient with malignant trophoblastic tumor
  Interventions: Drug: Toripalimab + ScTIL

INTERVENTIONS:
Drug: Toripalimab + ScTIL — Toripalimab (80 mg iv) 24 hours before or concomitantly with ScTIL 3-5x10^9 intravenous reinfusion.

SUMMARY:
The purpose of this study is to evaluate the safety and clinical efficacy of ScTIL in the treatment of recurrent or refractory cervical cancer, ovarian cancer and malignant trophoblastic tumor, to evaluate the pharmacokinetic characteristics of ScTIL, and to explore and analyze the changes of CTC, ctDNA and immunohistochemical Library of malignant tumor subjects before and after ScTIL treatment.Treatment will be terminated upon progressive disease, unacceptable toxicity, or withdrawal of consent. Subjects with responses other than progressive disease will receive subsequent rounds of ScTIL treatment.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and clinical efficacy of ScTIL in the treatment of recurrent or refractory cervical cancer, ovarian cancer and malignant trophoblastic tumor, to evaluate the pharmacokinetic characteristics of ScTIL, and to explore and analyze the changes of CTC, ctDNA and immunohistochemical Library of malignant tumor subjects before and after ScTIL treatment. Treatment will be terminated upon progressive disease, unacceptable toxicity, or withdrawal of consent. Subjects with responses other than progressive disease will receive subsequent rounds of ScTIL treatment.

The primary endpoint was objective response rate, defined as the proportion of patients with complete or partial response. Secondary endpoints were duration of response (time from the first evidence of response to disease progression or death, whichever came first), progression-free survival (time from the treatment initiation to disease progression or death, whichever came first), overall survival (time from the treatment initiation to the date of death or end of follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75, female;
2. Expected survival time > 3 months;
3. Clinically diagnosed advanced gynecological tumors, including:

   1. cervical cancer;
   2. Ovarian cancer;
   3. Malignant trophoblastic tumor;
4. Patients who have received radical surgery ± adjuvant radiotherapy and chemotherapy, or who have disease progression or recurrence after receiving too many lines of radiotherapy and chemotherapy, who have been unable to be resected again or who cannot tolerate radiotherapy and chemotherapy;
5. Patients with cervical and ovarian cancer have at least one measurable lesion according to RECIST version 1.1 standard; Patients with malignant trophoblastic tumor β HCG ≥ 5, with or without measurable lesions.
6. Voluntarily accept peripheral blood apheresis ± surgical resection of fresh tumor tissue to obtain cells for cell preparation, and the proportion of peripheral blood PD-1 positive T cells in the total T cells is ≥ 18%. For patients who have received PD-1 monoclonal antibody treatment before screening, the proportion of peripheral blood PD1 positive T cells in the total T cells is ≥ 10%;
7. The ECOG physical condition score is 0 to 1;
8. Have sufficient bone marrow and organ functions:

   Blood system (no blood transfusion or hematopoietic stimulating factor treatment within 14 days):

   Neutrophil count (ANC) ≥ 1.5 × one hundred and nine Platelet (PLT) ≥ 75 × 109/L Hemoglobin (HB) ≥ 90g / L Lymphocyte count (lym) ≥ 60% of the lower limit of normal value Lymphocyte subsets: proportion of B lymphocytes (CD19 +) in lymphocytes ≥ lower limit of normal value

   Liver function:

   Total bilirubin (TBIL) ≤ 1.5 × ULN Alanine aminotransferase (ALT) ≤ 3 × ULN Patients with liver metastasis or liver cancer: ≤ 5 × ULN Aspartic acid amino transfer (AST) ≤ 3 × ULN Patients with liver metastasis or liver cancer: ≤ 5 × ULN

   Renal function Creatinine ≤ 1.5 × ULN Coagulation function Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN International normalized ratio (INR) ≤ 1.5 × ULN
9. Fertile women must agree to permanently use reliable contraceptive methods (hormone or barrier method or abstinence, etc.) with their partners during and after the trial; Women of childbearing age (as defined in Appendix 9) must have a negative blood or urine pregnancy test within 7 days before the first use of the study drug;
10. The subjects must be informed of the study before the test and voluntarily sign a written informed consent.

Exclusion Criteria:

1. Central nervous system metastasis or meningeal metastasis with clinical symptoms, or there is other evidence that the patient's central nervous system metastasis or meningeal metastasis has not been controlled, which is not suitable for inclusion according to the judgment of the researcher;
2. Subjects with a history of second malignancy within 5 years before signing the informed consent;
3. Patients who had previously received PD-L1 mAb;
4. Those who have active infection within 1 week before apheresis and currently need systematic anti infection treatment;
5. Received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy, traditional Chinese medicine with anti-tumor indications and other anti-tumor treatments within 2 weeks before apheresis, Except for the following:

   1. Nitrosourea or mitomycin C were within 6 weeks before single harvest;
   2. Oral fluorouracils and small molecule targeted drugs were taken 1 week before apheresis.
6. Within 2 weeks before apheresis:

   1. Have received systemic glucocorticoid (prednisone > 10mg/day or equivalent dose of similar drugs) or other immunosuppressant treatment; Except for the following cases: local, eye, intra-articular, intranasal and inhaled glucocorticoids; Short term use of glucocorticoids for preventive treatment (e.g. prevention of contrast agent allergy);
   2. Used immunomodulatory drugs, including but not limited to thymosin, interleukin-2, interferon, etc;
7. Within 4 weeks before apheresis:

   1. Have received other unlisted clinical research drugs or treatments;
   2. Have undergone major organ surgery (excluding puncture biopsy) or significant trauma, or need to undergo elective surgery during the trial;
   3. Used live attenuated vaccine;
8. Currently suffering from interstitial lung disease;
9. Had received PD-1 monoclonal antibody treatment and had ≥ grade 2 Irae; Or other immunotherapy with ≥ grade 3 Irae;
10. Patients with active, or had, and relapsed autoimmune diseases, such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc., except for clinically stable autoimmune thyroid disease and well controlled type I diabetes.
11. The adverse reactions of previous anti-tumor treatment have not recovered to CTCAE 5.0 and the evaluation is ≤ 1 (except for the toxicity without safety risk judged by the researchers such as hair loss).
12. Have a history of immune deficiency, including HIV antibody test positive;
13. Hepatitis B: the titer of HBsAg (+) and/or hepatitis B DNA is higher than that of the research center. And/or hepatitis C: anti HCV positive; And/or Treponema pallidum antibody positive;
14. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    1. There are serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, ⅱ-ⅲ degree atrioventricular block, etc.
    2. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other grade 3 and above cardiovascular events occurred within 6 months before the first administration.
    3. New York Heart Association (NYHA) cardiac function grade ≥ grade II or left ventricular ejection fraction (LVEF) < 50%, or structural heart disease with high risk judged by other researchers;
    4. Clinically uncontrollable hypertension.
15. Serous effusion beyond clinical control is not suitable to be included in the group according to the judgment of the researcher;
16. Known alcohol or drug dependence;
17. Mental disorder or poor compliance;
18. Women with reproductive needs and pregnant or lactating women;
19. There are other serious or uncontrolled systemic diseases, or other reasons that are not suitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2022-04-18 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 12 weeks
  The proportion of patients with complete or partial response of cervical and ovarian cancer according to RECIST version 1.1, malignant trophoblastic tumor according to serum hCG level. Complete response was defined as a normal hCG level measured for 3 consecutive weeks. Partial response was defined as a ≥50% decrease in hCG level from baseline after 2 cycles.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 12 weeks
  The percentage of cases with remission and stable lesions after treatment in the total number of evaluable cases.
Duration of response (DOR) | 12 weeks
  The time from the first evidence of response to disease progression or death, whichever comes first.
Progression-free survival | 12 weeks
  The time from the treatment initiation to disease progression or death, whichever comes first.
Overall survival | 12 weeks
  The time from the treatment initiation to the date of death or end of follow-up.

IPD SHARING:
Plan to Share IPD: No